CLINICAL TRIAL: NCT02392507
Title: A Single-Arm, Multicenter, Open-Label, Phase 2 Study of Nab®-Paclitaxel (Abraxane®) and Carboplatin Chemotherapy Plus Necitumumab (LY3012211) in the First-Line Treatment of Patients With Stage IV Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Nab-Paclitaxel and Carboplatin Plus Necitumumab (LY3012211) in Participants With Stage IV Squamous NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15529; I4X-MC-JFCP (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-03-16; First posted 2015-03-19 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2019-11-15

CONDITIONS: Carcinoma, Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — necitumumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Necitumumab + Nab-Paclitaxel + Carboplatin (Experimental): Induction: Necitumumab administered intravenously (IV) at 800 milligram (mg) on day 1 and 8 of each cycle (3 week cycles); nab-paclitaxel administered IV at 100 milligram per square meter (mg/m²) on day 1, 8 and 15 of each cycle; carboplatin administered IV at a concentration of AUC (area under curve) 6 milligram per milliliter over time (mg*min/mL) on day 1 of each cycle, for a maximum of 4 cycles.
  Maintenance: Necitumumab administered IV at 800 mg on day 1 and 8 of each cycle; nab-paclitaxel administered IV at 100mg/m² on day 1 and 8 of each cycle (3 week cycles).
  Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Necitumumab; Drug: Nab-Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Necitumumab — Administered IV
  Other Names: LY3012211; IMC-11F8
Drug: Nab-Paclitaxel — Administered IV
  Other Names: Abraxane
Drug: Carboplatin — Administered IV

SUMMARY:
The purpose of the study is to determine if nab-paclitaxel and carboplatin chemotherapy plus necitumumab is effective and safe in participants with stage IV squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed squamous NSCLC.
* Have stage IV disease at the time of study entry (American Joint Committee on Cancer [AJCC] Staging Manual, 7th edition).
* Have measurable disease at the time of study enrollment as defined by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1).
* Have tumor tissue available for biomarker analysis.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Have adequate organ functions.

Exclusion Criteria:

* Are currently enrolled in another clinical trial.
* Have received prior anticancer therapy with monoclonal antibodies, signal transduction inhibitors, or any therapies targeting the epidermal growth factor receptor (EGFR), vascular endothelial growth factor (VEGF), or VEGF receptor.
* Have received previous chemotherapy for advanced NSCLC. Participants who have received adjuvant or neoadjuvant chemotherapy are eligible if the last administration of the prior regimens occurred at least 1 year prior to study entry.
* Have undergone major surgery or received any investigational therapy in the 4 weeks prior to study entry.
* Have undergone systemic radiotherapy within 4 weeks prior to study entry, or focal radiotherapy within 2 weeks prior to study entry.
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required).
* Have a history of arterial or venous embolism within 6 months prior to study entry.
* Have clinical evidence of concomitant infectious conditions.
* Have a known allergy / history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab, or any other contraindication to one of the administered treatments.
* Are pregnant or breastfeeding.
* Have a known history of drug abuse.
* Have a concurrent active malignancy. Participants with a history of malignancy are eligible provided the participant has been disease-free for ≥3 years, with the following exception: Participants with adequately treated basal or squamous cell carcinoma of the skin, preinvasive carcinoma of the cervix, or any cancer that in the judgment of the investigator and Lilly clinical research physician/designee may not affect the interpretation of results (for example, prostate, bladder) are eligible.
* Have discontinued investigational product or non approved use of a drug or device from a clinical trial within 30 days before the first day of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Florida Hospital Cancer Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Click here for more information about this study: A Study of Nab-Paclitaxel and Carboplatin Plus Necitumumab (LY3012211) in Participants With Stage IV Squamous NSCLC — http://www.lillytrialguide.com/en-US/studies/non-small-cell%20lung%20cancer/JFCP#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with known best overall response and off study treatment were considered to be completed.
Period: Induction Regimen
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Started | 54
Received at Least 1 Dose of Study Drug | 54
Completed | 47
Not Completed | 7
Not completed — Death | 3
Not completed — On Study Treatment at Study Conclusion | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Period: Maintenance Regimen
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Started | 34 (After induction regimen participants with disease response are eligible for maintenance regimen.)
Completed | 32
Not Completed | 2
Not completed — Death | 1
Not completed — On Study Treatment at Study Conclusion | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Necitumumab + Nab-Paclitaxel + Carboplatin: Induction: Necitumumab administered IV at 800 mg on day 1 and 8 of each cycle (3 week cycles); nab-paclitaxel administered IV at 100 mg/m² on day 1, 8 and 15 of each cycle; carboplatin administered IV at a concentration of AUC 6 mg*min/mL on day 1 of each cycle, for a maximum of 4 cycles.
  Maintenance: Necitumumab administered IV at 800 mg on day 1 and 8 of each cycle; nab-paclitaxel administered IV at 100mg/m² on day 1 and 8 of each cycle (3 week cycles).
  Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.96 (7.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
  Germany | 4
  Spain | 27
  Greece | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response or Partial Response (Objective Tumor Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of nontarget lesions, and no appearance of new lesions. Progressive disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: From Date of Randomization to Objective Disease Progression (Up to 18 Months)
Population: All randomized participants who received at least 1 dose of study drug and who had a complete radiographic assessment at baseline and at least 1 complete radiographic assessment post-baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 51
percentage of participants | 51.0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as time from date of randomization until first radiographic documentation of measured PD defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. PD was at least 20% increase in sum of diameters of target lesions with reference being smallest sum on study and an absolute increase of at least 5 mm,or unequivocal progression of non-target lesions,or 1 or more new lesions.If participant does not have complete baseline disease assessment,PFS time censored at date of randomization,regardless of whether or not objectively determined disease progression or death observed for participant.If participant was not known to have died or have objective progression as of data inclusion cutoff date for analysis,the PFS time censored at last adequate tumor assessment date.The use of new anticancer therapy prior to occurrence of PD resulted in censoring at the date of last radiographic assessment prior to initiation of new therapy.
Time Frame: From Date of Randomization to Measured Progressive Disease or Death Due to Any Cause (Up to 18 Months)
Population: All randomized participants who received at least 1 dose of study drug. Censored participants = 15.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 54
Months | 5.59 [4.24 to 7.69]

3. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from the date of randomization to the date of death due to any cause. Participants who are alive at the time of study completion or are lost to follow-up will be censored at the time they were last known to be alive.
Time Frame: From Date of Randomization until Death Due to Any Cause (Up to 18 Months)
Population: All randomized participants who received at least 1 dose of study drug. Censored participants = 35.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 54
Months | 15.54 [10.18 to NA] — The upper limit of the 95% CI was not calculated due to the high censoring rate.

4. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Disease Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD) (Disease Control Rate [DCR])
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and nontarget lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: From Date of Randomization to Objective Disease Progression or Start of New Anticancer Therapy (Up to 18 Months)
Population: All randomized participants who received at least 1 dose of study drug and who had a complete radiographic assessment at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 51
percentage of participants | 78.4

5. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab, Nab-Paclitaxel, and Carboplatin
Description: The Cmin is the minimum observed serum/plasma concentration of Necitumumab, Nab-Paclitaxel, and Carboplatin.
Time Frame: Cycle 3 and cycle 4: predose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Necitumumab: Necitumumab administered IV at 800 mg on day 1 and 8 of each cycle (3 week cycles).
- Carboplatin: Carboplatin administered IV at a concentration of AUC 6 mg*min/mL on day 1 of each cycle, for a maximum of 4 cycles.
- Paclitaxel: Nab-paclitaxel administered IV at 100 mg/m² on day 1, 8 and 15 of each cycle.
Arm/Group | Necitumumab | Carboplatin | Paclitaxel
Number analyzed (Participants) | 37 | 32 | 3
nanogram per milliliter (ng/mL)
  Cycle 3: number analyzed (Participants) | 37 | 32 | 2
  Cycle 3 | 65.2 (86.9) | 0.131 (36) | 33.6 (393)
  Cycle 4: number analyzed (Participants) | 30 | 31 | 3
  Cycle 4 | 90 (74.9) | 0.209 (197) | 107 (313)

6. Secondary Outcome: PK: Maximum Concentration (Cmax) of Necitumumab, Nab-Paclitaxel, and Carboplatin
Description: The Cmax is the maximum observed serum/plasma concentration of Necitumumab, Nab-Paclitaxel, and Carboplatin.
Time Frame: Cycle 1, 3 and 4: predose and <15minutes (min) post end-of-infusion
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Necitumumab: Necitumumab administered IV 800 mg on day 1 and 8 of each cycle (3 week cycles).
Arm/Group | Necitumumab | Carboplatin | Paclitaxel
Number analyzed (Participants) | 36 | 32 | 37
ng/mL
  Cycle 1 | 231 (27.1) | 16.4 (22) | 343 (81.2)
  Cycle 3: number analyzed (Participants) | 30 | 27 | 31
  Cycle 3 | 291 (46.5) | 16 (26.4) | 284 (73)
  Cycle 4: number analyzed (Participants) | 29 | 29 | 30
  Cycle 4 | 277 (42.5) | 10.5 (160) | 221 (77.6)

7. Secondary Outcome: Immunogenicity: Number of Participants Developing Anti-drug Antibodies to Necitumumab
Description: A participant was considered to have an anti-drug antibody response if anti-drug antibodies (ADA) were detected at any time point.
Time Frame: Predose Cycle 1 Through Short Term Follow Up (Up To 18 Months)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data for antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Necitumumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 54
Participants | 3

ADVERSE EVENTS:
Time Frame: Baseline Up to 49 Months
Description: All randomized participants who received at least 1 dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Necitumumab + Nab-paclitaxel + Carboplatin: Induction Phase: Necitumumab administered IV at 800 mg on day 1 and 8 of each cycle (3 week cycles); nab-paclitaxel administered IV at 100 mg/m² on day 1, 8 and 15 of each cycle; carboplatin administered IV at a concentration of AUC 6 mg*min/mL on day 1 of each cycle, for a maximum of 4 cycles. Participants may continue to receive treatment until discontinuation criteria are met.
- Necitumumab + Nab-paclitaxel: Maintenance Phase: Necitumumab administered IV at 800 mg on day 1 and 8 of each cycle; nab-paclitaxel administered IV at 100mg/m² on day 1 and 8 of each cycle (3 week cycles). Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Necitumumab + Nab-paclitaxel + Carboplatin: Induction Phase | Necitumumab + Nab-paclitaxel: Maintenance Phase
All-Cause Mortality (participants affected / at risk) | 3/54 | 1/34
Serious Adverse Events (participants affected / at risk) | 18/54 | 5/34
Other Adverse Events (participants affected / at risk) | 54/54 | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab + Nab-paclitaxel + Carboplatin: Induction Phase (N=54) | Necitumumab + Nab-paclitaxel: Maintenance Phase (N=34)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Necitumumab + Nab-paclitaxel + Carboplatin: Induction Phase (N=54) | Necitumumab + Nab-paclitaxel: Maintenance Phase (N=34)
Anaemia (Blood and lymphatic system disorders) | 34 (101) | 15 (27)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (24) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 19 (36) | 4 (6)
Nausea (Gastrointestinal disorders) | 16 (25) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 7 (11) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (14) | 3 (3)
Asthenia (General disorders) | 8 (14) | 2 (2)
Fatigue (General disorders) | 32 (77) | 6 (10)
Mucosal inflammation (General disorders) | 3 (8) | 0 (0)
Oedema peripheral (General disorders) | 6 (6) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 3 (3)
Conjunctivitis (Infections and infestations) | 3 (4) | 1 (3)
Paronychia (Infections and infestations) | 2 (2) | 5 (9)
Respiratory tract infection (Infections and infestations) | 9 (12) | 6 (8)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Vaginal infection (Infections and infestations) | 1/12 (1) | 0/6 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 6 (8) | 2 (3)
Lymphocyte count decreased (Investigations) | 6 (22) | 6 (11)
Neutrophil count decreased (Investigations) | 32 (85) | 1 (1)
Platelet count decreased (Investigations) | 17 (38) | 2 (2)
Weight decreased (Investigations) | 5 (5) | 0 (0)
White blood cell count decreased (Investigations) | 12 (46) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 13 (22) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (21) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (16) | 1 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (14) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 26 (60) | 7 (25)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (9) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 12 (27) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 5 (6) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (6)
Peripheral motor neuropathy (Nervous system disorders) | 4 (6) | 2 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9) | 9 (17)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 1 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 16 (32) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (11) | 5 (5)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 20 (59) | 6 (9)
Skin fissures (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-09-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT02392507/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT02392507/SAP_001.pdf